CLINICAL TRIAL: NCT04568434
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of AKCEA-APOCIII-LRx Administered Subcutaneously to Patients With Familial Chylomicronemia Syndrome (FCS)
Brief Title: A Study of Olezarsen (Formerly Known as AKCEA-APOCIII-LRx) Administered to Patients With Familial Chylomicronemia Syndrome (FCS)
Acronym: BALANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 678354-CS3; 2020-002536-67 (EudraCT Number)
Expanded Access: NCT06360237 (Approved for marketing)
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Familial Chylomicronemia Syndrome
Keywords: FCS
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome | interventions — olezarsen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants received olezarsen-matching placebo, once every 4 weeks by subcutaneous (SC) injection, during Weeks 1 to 49 of the 53-week treatment period.
  Interventions: Drug: Placebo
- Olezarsen 50 mg (Experimental): Participants received olezarsen, 50 milligrams (mg), once every 4 weeks by SC injection, during Weeks 1 to 49 of the 53-week treatment period.
  Interventions: Drug: Olezarsen
- Olezarsen 80 mg (Experimental): Participants received olezarsen 80 mg, once every 4 weeks by SC injection, during Weeks 1 to 49 of the 53-week treatment period.
  Interventions: Drug: Olezarsen

INTERVENTIONS:
Drug: Olezarsen — Olezarsen was administered by SC injection.
  Other Names: ISIS 678354; AKCEA-APOCIII-LRx
  Arms: Olezarsen 50 mg; Olezarsen 80 mg
Drug: Placebo — Olezarsen-matching placebo was administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of the study was to evaluate the efficacy of olezarsen as compared to placebo on the percent change in fasting triglycerides (TG) from baseline.

DETAILED DESCRIPTION:
This was a multi-center, double-blind, Phase 3 study in up to 60 patients with FCS. Participants were randomized in a 2:1 ratio to receive Olezarsen or matching placebo in a 53-week treatment period. The length of participation in the study was approximately 74 weeks, which included an up to 8-week screening period, a 53-week treatment period, and a 13-week post-treatment evaluation period. Following the treatment period, eligible patients had the option to enroll in the Open-label Extension (OLE) Study ISIS 678354-CS13 (NCT05130450).

ELIGIBILITY:
Key Inclusion Criteria:

* A diagnosis of genetically confirmed Familial Chylomicronemia Syndrome (type 1 Hyperlipoproteinemia)
* Fasting TG ≥ 880 mg/dL (10 millimoles per liter (mmol/L) at Screening
* History of pancreatitis. Patients without a documented history of pancreatitis are also eligible but their enrollment will be capped at 35%
* Stable doses of statins, omega-3 fatty acids, fibrates, or other lipid-lowering medications are allowed

Key Exclusion Criteria:

* Acute coronary syndrome within 6 months of Screening
* Major surgery within 3 months of Screening
* Have any other conditions, which, in the opinion of the Investigator would make the participant unsuitable for inclusion, or could interfere with participating in or completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (17):
  - Diabetes/Lipid Management & Research Center, Huntington Beach, California
  - University of California, San Francisco (UCSF) - Medical Center, San Francisco, California
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Advocate Health and Hospitals Corporation - Lutheran General Hospital, Park Ridge, Illinois
  - Ascension St. Vincent Cardiovascular Research Institute, Indianapolis, Indiana
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - University of Michigan- Endocrinology & Metabolism, Ann Arbor, Michigan
  - New York University (NYU) Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - York Clinical Research LLC, Norfolk, Virginia
  - West Virginia University Heart and Vascular Institute, Morgantown, West Virginia
- Canada (4):
  - Ecogene-21, Chicoutimi, Quebec
  - Nathalie Saint-Pierre, Montreal, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec, Quebec
  - Institute de Recherches Cliniques de Montreal, Montreal
- France (3):
  - Hôpital Louis Pradel - HCL, Bron
  - CHU Dijon - Bocage, Dijon
  - Assistance Publique - Hopitaux de Marseille, Marseille
- Italy (4):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
- Netherlands (3):
  - Academic Medical Center - Department of Vascular Medicine, Amsterdam
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- The Lipid Clinic (Oslo University Hospital), Oslo, Norway
- Portugal (3):
  - Centro Hospitalar de Lisboa Ocidental. E.P.E, - Hospital Santa Cruz, Carnaxide
  - Hospital da Senhora da Oliveira - Guimaraes, Creixomil
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
- Metabolicke centrum MUDr Katariny Raslovej s. r. o., Bratislava, Slovakia
- Spain (5):
  - Hospital Abente y Lago, A Coruña
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Fundacio Pere Virgili, Tarragona
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Solna
- United Kingdom (4):
  - The Royal Free Hospital, London
  - St. Thomas' Hospital, London
  - Manchester University NHS Foundation Trust (MFT), Manchester
  - Sandwell General Hospital, West Bromwich

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/

REFERENCES:
- [Result] Stroes ESG, Alexander VJ, Karwatowska-Prokopczuk E, Hegele RA, Arca M, Ballantyne CM, Soran H, Prohaska TA, Xia S, Ginsberg HN, Witztum JL, Tsimikas S; Balance Investigators. Olezarsen, Acute Pancreatitis, and Familial Chylomicronemia Syndrome. N Engl J Med. 2024 May 16;390(19):1781-1792. doi: 10.1056/NEJMoa2400201. Epub 2024 Apr 7. PMID 38587247
- [Derived] Sikora Kessler A, Vera-Llonch M, Karwatowska-Prokopczuk E, Alexander VJ, Ann Q, Mejia Herrera C, Paparrodopoulos S, Xia S, Stroes ESG, Baum SJ, Tsimikas S; Balance Investigators. Olezarsen reduces all-cause health services utilization and improves the treatment experience of patients with familial chylomicronemia syndrome. J Clin Lipidol. 2025 Dec 19:S1933-2874(25)00547-1. doi: 10.1016/j.jacl.2025.12.018. Online ahead of print. PMID 41545246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigative sites in the United States, Canada, France, Italy, Netherlands, Norway, Portugal, Slovakia, Spain, Sweden and the United Kingdom from 18 November 2020 to 17 October 2023.
Pre-assignment Details: Participants with Familial Chylomicronemia Syndrome (FCS) were enrolled and randomized to receive either olezarsen (50 milligrams [mg] or 80 mg) or olezarsen-matching placebo for a 53-week treatment period. Participants completing treatment had an option to enroll in the Open-label Extension (OLE) Study ISIS 678354-CS13 (NCT05130450).
Groups:
- Placebo: Participants received olezarsen-matching placebo, once every 4 weeks by SC injection, during Weeks 1 to 49 of the 53-week treatment period.
- Olezarsen 50 mg: Participants received olezarsen 50 mg, once every 4 weeks by SC injection, during Weeks 1 to 49 of the 53-week treatment period.
Period: Overall Study
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Started | 23 | 21 | 22
Completed | 22 | 19 | 19
Not Completed | 1 | 2 | 3
Not completed — Voluntary Withdrawal | 0 | 1 | 1
Not completed — Adverse Events (AE) or Serious Adverse Events (SAE) | 0 | 1 | 2
Not completed — Investigator Judgement | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants that were randomly assigned to treatment and received at least 1 dose of olezarsen or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg | Total
Number analyzed (Participants) | 23 | 21 | 22 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (14.67) | 43.2 (12.11) | 47.7 (13.30) | 45 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 11 | 38
  Male | 11 | 6 | 11 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 1 | 7
  Not Hispanic or Latino | 20 | 18 | 21 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 22 | 17 | 17 | 56
  More than one race | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Fasting Triglycerides (TG) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 2595.7 (1255.72) | 2683.8 (1235.06) | 2613.1 (1498.96) | 2629.5 (1315.45)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting TG at Month 6
Time Frame: Baseline, Month 6
Population: FAS included all participants that were randomly assigned to treatment and received at least 1 dose of olezarsen or placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Number analyzed (Participants) | 23 | 21 | 22
percent change | 11.52 [-5.321 to 28.356] | -10.85 [-27.797 to 6.095] | -31.99 [-49.031 to -14.940]
Statistical Analysis 1: Comparison: Placebo vs Olezarsen 80 mg; Test type: Superiority; p = 0.0009, ANCOVA — ANCOVA model included effects of treatment (olezarsen 80 mg, olezarsen 50 mg, or placebo): dependent variable, protocol specified 2 randomization stratification factors: fixed effects, log-transformed baseline TG: covariate; LS mean difference = -43.5, 95% CI 2-sided [-69.085 to -17.921]
Statistical Analysis 2: Comparison: Placebo vs Olezarsen 50 mg; Test type: Superiority; p = 0.0775, ANCOVA — Analysis of covariance (ANCOVA) model included effects of treatment (olezarsen 80 mg, olezarsen 50 mg, or placebo): dependent variable, protocol specified 2 randomization stratification factors: fixed effects, log-transformed baseline TG: covariate; Least squares (LS) mean difference = -22.37, 95% CI 2-sided [-47.200 to 2.463]

2. Secondary Outcome: Percent Change From Baseline in Fasting TG at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Number analyzed (Participants) | 23 | 21 | 22
percent change | 20.89 [1.016 to 40.764] | -22.92 [-42.505 to -3.336] | -38.50 [-58.187 to -18.815]
Statistical Analysis 1: Comparison: Placebo vs Olezarsen 50 mg; Test type: Superiority; p = 0.0044, ANCOVA — ANCOVA model included percent change from baseline in fasting TG at Month 12: dependent variable, treatment group, protocol specified 2 randomization stratification factors: fixed effects, log-transformed baseline TG: covariate; LS mean difference = -43.81, 95% CI 2-sided [-73.928 to -13.692]
Statistical Analysis 2: Comparison: Placebo vs Olezarsen 80 mg; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = -59.39, 95% CI 2-sided [-90.663 to -28.119]

3. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein C-III (apoC-III) at Months 6 and 12
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Number analyzed (Participants) | 23 | 21 | 22
percent change
  Month 6 | 7.57 [-5.229 to 20.359] | -57.91 [-71.193 to -44.631] | -66.13 [-79.437 to -52.823]
  Month 12 | 17.08 [2.149 to 32.009] | -59.98 [-75.163 to -44.795] | -64.20 [-79.408 to -48.984]
Statistical Analysis 1: Comparison: Placebo vs Olezarsen 50 mg; Percent Change from Baseline at Month 6; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model included percent change from baseline in fasting apoC-III at Month 6: dependent variable, treatment group, protocol specified 2 randomization stratification factors: fixed effects, log-transformed baseline apoC-III: covariate; LS mean difference = -65.48, 95% CI 2-sided [-82.634 to -48.320]
Statistical Analysis 2: Comparison: Placebo vs Olezarsen 80 mg; Percent Change from Baseline at Month 6; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -73.69, 95% CI 2-sided [-94.553 to -52.837]
Statistical Analysis 3: Comparison: Placebo vs Olezarsen 50 mg; Percent Change from Baseline at Month 12; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model included percent change from baseline in fasting apoC-III at Month 12: dependent variable, treatment group, protocol specified 2 randomization stratification factors: fixed effects, log-transformed baseline apoC-III: covariate; Ls mean difference = -77.06, 95% CI 2-sided [-98.938 to -55.177]
Statistical Analysis 4: Comparison: Placebo vs Olezarsen 80 mg; Percent Change from Baseline at Month 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 3]; LS mean difference = -81.28, 95% CI 2-sided [-104.656 to -57.894]

4. Secondary Outcome: Percentage of Participants With ≥ 40% Reduction in Fasting TG at Month 6
Description: Percentages are rounded off to the nearest single decimal place.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Number analyzed (Participants) | 23 | 21 | 22
percentage of participants | 4.3 | 33.3 | 40.9

5. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein B-48 (apoB-48) at Months 6 and 12
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Number analyzed (Participants) | 23 | 21 | 22
percent change
  Month 6 | 24.50 [-9.972 to 58.973] | -8.78 [-42.976 to 25.406] | -59.46 [-93.164 to -25.765]
  Month 12 | -3.52 [-53.159 to 46.124] | -36.41 [-77.689 to 4.860] | -79.15 [-118.442 to -39.861]
Statistical Analysis 1: Comparison: Placebo vs Olezarsen 50 mg; Percent Change From Baseline at Month 6; Test type: Superiority; p = 0.1860, ANCOVA — ANCOVA model included percent change from baseline in fasting apoB-48 to Month 6: dependent variable, treatment group, protocol prespecified randomization stratification factors: fixed effects & log-transformed baseline apoB-48: covariate; LS mean difference = -33.29, 95% CI 2-sided [-82.612 to 16.041]
Statistical Analysis 2: Comparison: Placebo vs Olezarsen 80 mg; Percent Change From Baseline at Month 6; Test type: Superiority; p = 0.0019, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -83.97, 95% CI 2-sided [-136.949 to -30.982]
Statistical Analysis 3: Comparison: Placebo vs Olezarsen 50 mg; Percent Change from Baseline at Month 12; Test type: Superiority; p = 0.4219, ANCOVA — ANCOVA model included percent change from baseline in fasting apoB-48 to Month 12: dependent variable, treatment group, protocol prespecified randomization stratification factors: fixed effects & log-transformed baseline apoB-48: covariate; LS mean difference = -32.9, 95% CI 2-sided [-113.254 to 47.459]
Statistical Analysis 4: Comparison: Placebo vs Olezarsen 80 mg; Percent Change from Baseline at Month 12; Test type: Superiority; p = 0.0560, ANCOVA — [p-value comment as in outcome 5, analysis 3]; LS mean difference = -75.63, 95% CI 2-sided [-153.195 to 1.927]

6. Secondary Outcome: Percent Change From Baseline in Fasting Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Months 6 and 12
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Number analyzed (Participants) | 23 | 21 | 22
percent change
  Month 6 | 5.33 [-5.345 to 16.014] | -12.35 [-23.541 to -1.163] | -18.86 [-29.952 to -7.774]
  Month 12 | 12.01 [-2.480 to 26.494] | -17.84 [-32.128 to -3.545] | -27.69 [-41.722 to -13.664]
Statistical Analysis 1: Comparison: Placebo vs Olezarsen 50 mg; Percent Change from Baseline Month 6; Test type: Superiority; p = 0.0401, ANCOVA — ANCOVA model included percent change from baseline in fasting non-HDL-C to Month 6: dependent variable, treatment group, protocol prespecified randomization stratification factors: fixed effects & log-transformed baseline non-HDL-C: covariate; LS mean difference = -17.69, 95% CI 2-sided [-34.571 to -0.801]
Statistical Analysis 2: Comparison: Placebo vs Olezarsen 80 mg; Percent Change from Baseline Month 6; Test type: Superiority; p = 0.0036, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference = -24.2, 95% CI 2-sided [-40.484 to -7.911]
Statistical Analysis 3: Comparison: Placebo vs Olezarsen 50 mg; Percent Change from Baseline at Month 12; Test type: Superiority; p = 0.0134, ANCOVA — ANCOVA model included percent change from baseline in fasting non-HDL-C to Month 12: dependent variable, treatment group, protocol prespecified randomization stratification factors: fixed effects & log-transformed baseline non-HDL-C: covariate; LS mean difference = -29.84, 95% CI 2-sided [-53.490 to -6.198]
Statistical Analysis 4: Comparison: Placebo vs Olezarsen 80 mg; Percent Change from Baseline at Month 12; Test type: Superiority; p = 0.0009, ANCOVA — [p-value comment as in outcome 6, analysis 3]; LS mean difference = -39.7, 95% CI 2-sided [-63.108 to -16.292]

7. Secondary Outcome: Adjudicated Acute Pancreatitis Mean Event Rate Per 100 Participant-Years During the Treatment Period (Week 1 Through Week 53) in Participants With Prior History of Pancreatitis
Description: All AEs and SAEs that consistently occurred during the study with an event of acute pancreatitis were adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis as outlined in the Acute Pancreatitis Adjudication Committee (PAC) Charter. These events were categorized as 1) documented pancreatitis, 2) probable pancreatitis, 3) possible pancreatitis, 4) unable to adjudicate and 5) no diagnosis of acute pancreatitis. The adjudicated event rate represents the average number of events per 100 participant-years during the treatment period.
Time Frame: During the treatment period Week 1 through Week 53
Population: FAS included all participants that were randomly assigned to treatment and received at least 1 dose of olezarsen or placebo. Overall number of participants analyzed is the number of participants with a history of pancreatitis within 10 years prior to screening. As prespecified in the protocol, data for this outcome measure was collected and reported in a pooled manner for olezarsen (combined Olezarsen 50 mg + Olezarsen 80 mg)
Measure: Mean (95% Confidence Interval); unit: events per 100 participant-years
Groups:
- Pooled Olezarsen: Participants received olezarsen 50 mg or 80 mg, once every 4 weeks by SC injection, during Weeks 1 to 49 of the 53-week treatment period.
Arm/Group | Placebo | Pooled Olezarsen
Number analyzed (Participants) | 15 | 32
events per 100 participant-years | 66.22 [30.490 to 143.817] | 6.73 [1.612 to 28.087]
Statistical Analysis 1: Comparison: Placebo vs Pooled Olezarsen; Test type: Superiority; p = 0.0052, Negative Binomial Regression Model — Regression model: treatment group & previous treatment (volanesorsen):factors adjudicated acute pancreatitis events in 5 years prior enrollment:covariate. Logarithm of time in year that each participant was observed from Week 1 to 53:offset variable; Mean Rate Ratio = 0.1, 95% CI 2-sided [0.020 to 0.506]

8. Secondary Outcome: Adjudicated Acute Pancreatitis Mean Event Rate Per 100 Participant-Years During the Treatment Period (Week 1 Through Week 53)
Description: All AEs and SAEs that consistently occurred during the study with an event of acute pancreatitis were adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis as outlined in the PAC Charter. These events were categorized as 1) documented pancreatitis, 2) probable pancreatitis, 3) possible pancreatitis, 4) unable to adjudicate and 5) no diagnosis of acute pancreatitis. The adjudicated event rate represents the average number of events per 100 participant-years during the treatment period.
Time Frame: During the treatment period Week 1 through Week 53
Population: FAS included all participants that were randomly assigned to treatment and received at least 1 dose of olezarsen or placebo. As prespecified in the protocol, data for this outcome measure was collected and reported in a pooled manner for olezarsen (combined Olezarsen 50 mg + Olezarsen 80 mg).
Measure: Mean (95% Confidence Interval); unit: events per 100 participant-years
Arm/Group | Placebo | Pooled Olezarsen
Number analyzed (Participants) | 23 | 43
events per 100 participant-years | 36.31 [14.700 to 89.685] | 4.37 [0.942 to 20.298]
Statistical Analysis 1: Comparison: Placebo vs Pooled Olezarsen; Test type: Superiority; p = 0.0144, Negative Binomial Regression Model — [p-value comment as in outcome 7, analysis 1]; Mean Rate Ratio = 0.12, 95% CI 2-sided [0.022 to 0.656]

9. Secondary Outcome: Adjudicated Acute Pancreatitis Mean Event Per 100 Participant-Years Rate During Week 13 Through Week 53 in Participants With Prior History of Pancreatitis
Description: All AEs and SAEs that consistently occurred during the study with an event of acute pancreatitis were adjudicated by a blinded, independent committee according to the Atlanta classification of acute pancreatitis as outlined in the PAC Charter. These events were categorized as 1) documented pancreatitis, 2) probable pancreatitis, 3) possible pancreatitis, 4) unable to adjudicate and 5) no diagnosis of acute pancreatitis. The adjudicated event rate represents the average number of events per 100 participant-years during the specified duration.
Time Frame: Week 13 through Week 53
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: events per 100 participant-years
Arm/Group | Placebo | Pooled Olezarsen
Number analyzed (Participants) | 15 | 32
events per 100 participant-years | 57.89 [24.469 to 136.972] | 8.17 [1.952 to 34.177]
Statistical Analysis 1: Comparison: Placebo vs Pooled Olezarsen; Test type: Superiority; p = 0.0174, Negative Binomial Regression Model — Regression model: treatment group & previous treatment (volanesorsen):factors adjudicated acute pancreatitis events in 5 years prior enrollment:covariate. Logarithm of time in year that each participant was observed from Week 13 to 53:offset variable; Mean Rate Ratio = 0.14, 95% CI 2-sided [0.028 to 0.709]

10. Secondary Outcome: Adjudicated Acute Pancreatitis Mean Event Rate Per 100 Participant-Years During Week 13 to Week 53
Description: as for outcome 9
Time Frame: Week 13 through Week 53
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: events per 100 participant-years
Arm/Group | Placebo | Pooled Olezarsen
Number analyzed (Participants) | 23 | 43
events per 100 participant-years | 33.43 [13.250 to 84.321] | 5.42 [1.229 to 23.897]
Statistical Analysis 1: Comparison: Placebo vs Pooled Olezarsen; Test type: Superiority; p = 0.0314, Negative Binomial Regression Model — [p-value comment as in outcome 9, analysis 1]; Mean Rate Ratio = 0.16, 95% CI 2-sided [0.031 to 0.850]

11. Secondary Outcome: Percentage of Participants With ≥ 70% Reduction in Fasting TG at Month 6
Description: Percentages are rounded off to the nearest single decimal place.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Number analyzed (Participants) | 23 | 21 | 22
percentage of participants | 0 | 4.8 | 9.1

12. Secondary Outcome: Percentage of Participants With Fasting TG ≤ 880 mg/dL at Month 6
Description: Percentages are rounded off to the nearest single decimal place.
Time Frame: Month 6
Population: FAS included all participants that were randomly assigned to treatment and received at least 1 dose of olezarsen or placebo. "Overall number of participants analyzed" indicates the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Number analyzed (Participants) | 21 | 20 | 21
percentage of participants | 0 | 10.0 | 14.3

13. Secondary Outcome: Adjudicated Acute Pancreatitis Mean Event Rate Per 100 Participant-Years During Treatment Period in Participants With ≥ 2 Events in 5 Years Prior to Enrollment
Description: as for outcome 8
Time Frame: During the treatment period Week 1 through Week 53
Population: FAS included all participants that were randomly assigned to treatment and received at least 1 dose of olezarsen or placebo. Overall number of participants analyzed is the number of participants with ≥ 2 adjudicated acute pancreatitis events in 5 years prior to enrollment. As prespecified in the protocol, data for this outcome measure was collected and reported in a pooled manner for olezarsen (combined Olezarsen 50 mg + Olezarsen 80 mg).
Measure: Mean (95% Confidence Interval); unit: events per 100 participant-years
Arm/Group | Placebo | Pooled Olezarsen
Number analyzed (Participants) | 9 | 12
events per 100 participant-years | 118.59 [61.226 to 229.698] | 16.59 [4.051 to 67.948]
Statistical Analysis 1: Comparison: Placebo vs Pooled Olezarsen; Test type: Superiority; p = 0.0137, Negative Binomial Regression Model — [p-value comment as in outcome 7, analysis 1]; Mean Rate Ratio = 0.14, 95% CI 2-sided [0.029 to 0.669]

14. Secondary Outcome: Adjudicated Acute Pancreatitis Mean Event Rate Per 100 Participant-Years From Week 13 to Week 53 in Participants With ≥ 2 Events in 5 Years Prior to Enrollment
Description: as for outcome 9
Time Frame: Week 13 to Week 53
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: events per 100 participant-years
Groups:
- Pooled Olezarsen: Participants received olezarsen 50 mg or 80 mg, once every 4 weeks by SC injection during Weeks 1 to 49 of the 53-week treatment period.
Arm/Group | Placebo | Pooled Olezarsen
Number analyzed (Participants) | 9 | 12
events per 100 participant-years | 106.91 [50.204 to 227.682] | 21.36 [5.233 to 87.219]
Statistical Analysis 1: Comparison: Placebo vs Pooled Olezarsen; Test type: Superiority; p = 0.0480, Negative Binomial Regression Model — Regression model:treatment group & previous treatment (volanesorsen):factors adjudicated acute pancreatitis events in 5 years prior enrollment:covariate. Logarithm of time in year that each participant was observed from Week 13 to 53:offset variable; Mean Rate Ratio = 0.2, 95% CI 2-sided [0.040 to 0.986]

15. Secondary Outcome: Percentage of Participants With Fasting TG ≤ 500 mg/dL at Month 6
Description: Percentages are rounded off to the nearest single decimal place.
Time Frame: Month 6
Population: FAS included all participants that were randomly assigned to treatment and received at least 1 dose of olezarsen or placebo. 'Overall number of participants analyzed' indicates the number of participants with data available for the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
Number analyzed (Participants) | 22 | 21 | 22
percentage of participants | 0 | 0 | 13.6

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to end of the follow-up (up to Week 66)
Description: Safety analysis set included all subjects that were randomly assigned to treatment and received at least 1 dose of olezarsen or placebo.
Arm/Group | Placebo | Olezarsen 50 mg | Olezarsen 80 mg
All-Cause Mortality (participants affected / at risk) | 0/23 | 1/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 9/23 | 4/21 | 3/22
Other Adverse Events (participants affected / at risk) | 19/23 | 17/21 | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Olezarsen 50 mg (N=21) | Olezarsen 80 mg (N=22)
Gastric varices (Gastrointestinal disorders) | 1 | 0 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 4 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 3 | 0 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 2 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pancreatogenous diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Olezarsen 50 mg (N=21) | Olezarsen 80 mg (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 2
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Fatigue (General disorders) | 4 | 1 | 1
Injection site erythema (General disorders) | 1 | 1 | 2
Injection site pain (General disorders) | 0 | 2 | 1
COVID-19 (Infections and infestations) | 8 | 6 | 3
Cellulitis (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 2 | 3 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 1 | 1
Platelet count decreased (Investigations) | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Headache (Nervous system disorders) | 3 | 4 | 1
Migraine (Nervous system disorders) | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT04568434/Prot_SAP_000.pdf